CLINICAL TRIAL: NCT04137302
Title: Administration of Hydrocortisone in Young Healthy Male Volunteers: Determination of Biomarkers for Distinguishing Between Local and Systemic Pathways
Brief Title: Administration of Hydrocortisone in Young Healthy Male Volunteers
Acronym: H-CORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Collaborators: French Anti-Doping Agency (AFLD) (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHRO 2019-04
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Anti-doping Campaign, Detection of Hydrocortisone
Keywords: Hydrocortisone (cortisol); local administration of cortisol; systemic administration of cortisol; biomarkers

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, open-label study
  Distribution of patients in groups according to a ratio (1:1)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical hydrocortisone administration (Active Comparator): dermal cream (twice a day, 2.5 g of cream, 1% hydrocortisone during 5 days)
  Interventions: Drug: Hydrocortisone administration
- Systemic hydrocortisone administration (Active Comparator): tablets (once a day, 50 mg, morning, during 50 days)
  Interventions: Drug: Hydrocortisone administration

INTERVENTIONS:
Drug: Hydrocortisone administration — Hydrocortisone administration with collection of blood, urine and saliva samples before (1 week), during (5 days) and after (1 week) the 2 treatments

SUMMARY:
The misuse of cortisone or hydrocortisone for doping purpose in sport has been widely reported in the literature, but to date, no formal testing procedure is available and applicable in an anti-doping laboratory to detect hydrocortisone doping abuse , i.e., administration by systemic way.

The investigators therefore propose to identify biomarkers that clearly distinguish between an authorized local administration of hydrocortisone and a prohibited systemic administration, by studying the impact of 5-day administration of hydrocortisone per 2 different routes.

DETAILED DESCRIPTION:
Clinical research with two groups of ten volunteers one group with 5 days with local administration (cream, applied to healthy skin) one group with 5 days with systemic route of administration (per os)

ELIGIBILITY:
Inclusion Criteria:

* male subjects

  * aged 18 to 30 years
  * 18 < BMI < 28
  * participating in regular physical activity (3-5 times/week)
  * subjects not on medication

Exclusion Criteria:

asthmatic subjects or history of respiratory or cardiac pathology; use of corticosteroids in the past 6 months; high blood pressure; ulcerated lesions of the skin, acne, rosacea; Infectious state (bacterial, viral, and fungal infections); diabetic subjects; ulcerative history and other gastrointestinal disorders; lactose allergy; galactose intolerance; ulcerative colonic pathology; myastenia gravis; live vaccine kidney failure

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Urinary concentration of cortisol and its metabolites with Gas Chromatography Mass Spectrometry | 7 days
  Gas Chromatography Mass Spectrometry to study biomarkers urine level at 8 am, 10 am, 8 pm
Urinary concentration of cortisol and its metabolites with Gas Chromatography Mass Spectrometry | Day 12
  Gas Chromatography Mass Spectrometry to study biomarkers urine level at 8 am,
Urinary concentration of cortisol and its metabolites with Isotope ratio mass spectrometry t | 7 days
  Isotope ratio mass spectrometry to study biomarkers urine level at 8 am, 10 am, 8 pm
Urinary concentration of cortisol and its metabolites with Isotope ratio mass spectrometry t | Day 12
  Isotope ratio mass spectrometry to study biomarkers urine level at 8 am

SECONDARY OUTCOMES:
blood concentration of cortisol | 7 days
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am; 10 am, 8 pm
blood concentration of cortisol | Day 12
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am;
blood concentration of DeHydroEpiAndrostérone | 7 days
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am; 10 am, 8 pm
blood concentration of DeHydroEpiAndrostérone | day 12
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am;
blood concentration of Adreno CorticoTrophic Hormone | 7 days
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am; 10 am, 8 pm
blood concentration of Adreno CorticoTrophic Hormone | Day 12
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am;
saliva concentration of cortisol | 7 days
  Elisa test (enzyme-linked immunosorbent assay, ) to study cortisol concentration at 8 am; 10 am, 8 pm
saliva concentration of DeHydroEpiAndrostérone | 7 days
  Elisa test (enzyme-linked immunosorbent assay, ) to study cortisol concentration at 8 am; 10 am, 8 pm
saliva concentration of Adreno CorticoTrophic Hormone | 7 days
  Elisa test (enzyme-linked immunosorbent assay, ) to study cortisol concentration at 8 am; 10 am, 8 pm
saliva concentration of cortisol | Day 12
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am
saliva concentration of Adreno CorticoTrophic Hormone | Day 12
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am
saliva concentration of DeHydroEpiAndrostérone | Day 12
  Elisa test (enzyme-linked immunosorbent assay) to study cortisol concentration at 8 am

CONTACTS AND LOCATIONS:
Overall Officials: AMIOT Virgile, MD, Study Director — Hospital Regional Center of ORLEANS
Locations (1):
- Regional Hospital Center of ORLEANS, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arlettaz A, Portier H, Lecoq AM, Rieth N, De Ceaurriz J, Collomp K. Effects of short-term prednisolone intake during submaximal exercise. Med Sci Sports Exerc. 2007 Sep;39(9):1672-8. doi: 10.1249/mss.0b013e3180dc992c. PMID 17805102
- [Background] Buisson C, Mongongu C, Frelat C, Jean-Baptiste M, de Ceaurriz J. Isotope ratio mass spectrometry analysis of the oxidation products of the main and minor metabolites of hydrocortisone and cortisone for antidoping controls. Steroids. 2009 Mar;74(3):393-7. doi: 10.1016/j.steroids.2008.11.001. Epub 2008 Nov 13. PMID 19056411
- [Background] Collomp K, Arlettaz A, Buisson C, Lecoq AM, Mongongu C. Glucocorticoid administration in athletes: Performance, metabolism and detection. Steroids. 2016 Nov;115:193-202. doi: 10.1016/j.steroids.2016.09.008. Epub 2016 Sep 16. PMID 27643452
- [Background] Collomp K, Arlettaz A, Portier H, Lecoq AM, Le Panse B, Rieth N, De Ceaurriz J. Short-term glucocorticoid intake combined with intense training on performance and hormonal responses. Br J Sports Med. 2008 Dec;42(12):983-8. doi: 10.1136/bjsm.2007.043083. Epub 2007 Nov 29. PMID 18048433